CLINICAL TRIAL: NCT00781118
Title: AngelMed for Early Recognition and Treatment of STEMI
Acronym: ALERTS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Angel Medical Systems (Industry)
Collaborators: Symbios Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ALERTS Study
Record Dates: First submitted 2008-10-24; First posted 2008-10-28 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Acute Myocardial Infarction (AMI); Coronary Occlusion; Acute Coronary Syndrome
Keywords: Acute Myocardial Infarction (MI); ST Shift; Coronary Occlusion; Acute Coronary Syndrome
MeSH Terms: conditions — Coronary Occlusion; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): The Treatment arm has alerting enabled in their device during the 6-month randomization period. Treatment arm patients also have alerting enabled in the post-randomization period. Once a patient arrives at the ER, the standard of care triage process for MI is followed and that is outside of the ALERTS Study protocol. With Amendment the Treatment arm was re-defined as an ALARMS_ON group which included A) Control patients after the randomization period and until database lock (4/1/2014); and, b) Treatment patients both during the randomization period and after the randomization period until database lock (4/1/2014).
  Interventions: Device: Guardian System
- Control (Other): The Control arm has alerting disabled in their device during the 6-month randomization period. Control arm patients also have alerting enabled in the post-randomization period. Once a patient arrives at the ER, the standard of care triage process for MI is followed and that is outside of the ALERTS Study protocol. With Amendment the Control arm was re-defined as an ALARMS_OFF group which included A) Control patients during the randomization period when the Guardian did not have alarms enabled.
  Interventions: Device: Guardian System

INTERVENTIONS:
Device: Guardian System — There is no intervention in this study. The device is a diagnostic only.

SUMMARY:
A prospective, randomized multicenter study of subjects with a high-risk of having a myocardial infarction (MI) due to acute coronary syndrome or bypass surgery. There is no differential intervention administered to the two arms of the ALERTS Study. The study evaluates whether or not a patient alarm from the Guardian System will provide benefit (e.g. shorten pre-hospital delay) compared to symptoms-only ER presentation in the event of a heart attack. An amendment to the data analysis protocol was collaboratively created by AngelMed and FDA, and was adopted by AngelMed on 4/22/2017.

DETAILED DESCRIPTION:
There are over one million acute myocardial infarctions (AMI) each year in the United States with more than 400,000 of these resulting in death. Early identification of AMI, and prompt treatment has been shown to significantly improve clinical outcomes. Experimental and clinical studies have shown that most of the irreversible damage to the myocardium occurs during the first two hours after coronary occlusion. Milavetz et al. demonstrated that successful reperfusion therapy within two hours was associated with the greatest degree of myocardial salvage. According to Boersma, et al., restoration of flow, regardless of the method used, can abort infarction within the first 30 minutes after coronary occlusion, and the benefit of fibrinolytic therapy compared with placebo is considerably higher in patients treated within 2 hours after symptom onset than in those treated later.2 Further, evidence exists that expeditious restoration of flow in the obstructed infarct artery after the onset of symptoms in patients with the most severe type of MI, ST elevation MI (STEMI) is a key determinant of short and long-term outcomes regardless of whether reperfusion is accomplished by fibrinolysis or percutaneous coronary intervention (PCI). Therefore, the early arrival at the hospital for a reliable diagnosis and initiation of treatment is paramount to improve the outcomes of myocardial infarction. However, despite efforts at educating the public over the past decade, the mean time from AMI symptom onset to arrival at a hospital for treatment has remained, disappointingly, at 2.5-3.0 hours.

The largest proportion of the total pre-hospital delay is the interval between the onset of symptoms and the decision to seek medical treatment. Finnegan et al. described that the reasons for delay in seeking medical evaluation generally stem from patient misconceptions about symptom experience, expectations, and attribution. In many cases, patients expect the type of heart attack that they often see in movies or on television: the kind of crushing chest pain that drops a person to the ground. The reality is that many heart attacks are much "quieter," causing only mild chest pain or discomfort or other symptoms such as shortness of breath or diaphoresis.

If patients would take action during the first hour following symptom onset, many lives and significant cost could be saved. It is technically possible to monitor EKGs and detect an acute infarction, even if the patient is unaware that he or she is experiencing a heart attack. However, currently available systems have limitations in the home environment. Twelve lead EKG systems require a clinically trained individual to place them. Holter monitors suffer from limitations in the ability to detect ST deviation due to low compliance and are limited in practice to 24 to 72 hours of monitoring. Systems using surface leads are all subject to noise and other artifacts from patient movement and body orientation, particularly if the patient is ambulatory.

A potentially ideal solution is to implant a device that measures heart signals from inside the heart and will alert the patient when it detects electrogram characteristics set by the physician as worthy of medical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Subject has at least one of the following conditions:

  1. Diabetes (Type I or Type II)
  2. Compromised renal function (Cr > 1.2 mg/dl or creatinine clearance less than 50)
  3. TIMI Risk Score ≥ 3
* Presents (within past 6 months) with a high-risk acute coronary syndrome (e.g., Unstable Angina, STEMI or NSTEMI) or has undergone or is scheduled for CABG within 6 months of implantation.
* Has already undergone coronary angiography and revascularization, unless the physician determines it is appropriate to implant before or during the planned procedure.
* Lives in a geographic area in close proximity (within 60 minutes by EMS) to any hospital that can treat AMI.
* Subjects (men or women) at least 21 years of age. Women of childbearing age must have a negative pregnancy test or confirmation of one of the following:

  1. Post-menopause or amenorrheic during the past year
  2. Surgical sterilization
  3. Use of effective contraceptive method

Exclusion Criteria:

* In the investigator's opinion, subject lacks ability to respond appropriately to alarms, e.g., illiteracy, poor memory or cognitive function, dementia or other condition affecting memory function, etc.
* There is known compromised tissue at the site of lead implantation in the apex of the right ventricle, e.g., prior infarct affecting the RV apex location.
* A permanent pacemaker or ICD is already in place or the patient is indicated for ICD or pacemaker implantation based on the guidelines published by the American College of Cardiology as Class I and IIa recommendations. Class IIb recommendations are at the investigator's discretion.
* Subject cannot feel the IMD vibration when placed on top of the skin on the left pectoral side of the chest.
* Subject has recurrent or persistent atrial fibrillation.
* Subject has recurrent or persistent non-sinus cardiac rhythm, second or third degree atrioventricular blocks, QRS duration greater than 120 ms, Benign Early Repolarization (BER), or Brugada Syndrome.
* Subject has left ventricular hypertrophy evidenced by EKG criteria.
* Subject has any condition preventing the subcutaneous implantation of the Guardian System in a left pectoral pouch, such as: superior vena cava thrombosis, subcutaneous tissue deemed inappropriate for the procedure or prior central venous access via portacath, Hickman, Groshong, or similar placed in a left pectoral location or left side PICC line.
* Subject has extremely heavy alcohol consumption (participates in binge drinking that leads to alcohol intoxication) or has history of alcohol or illicit drug abuse within past 5 years.
* There is evidence of unresolved infection (fever > 38° C and/or leukocytosis > 15,000).
* Subject has history of bleeding disorders or severe coagulopathy (platelets < 100,000 plts/ml; APTT or PT > 1.3 x reference range).
* Subject has had a hemorrhagic stroke or transient ischemic attack (TIA) in the past 6 months.
* Subject has other severe diseases, such as cancer or refractory congestive heart failure, associated with limitation of life expectancy (less than 1 year), which may lead to inadequate compliance to the protocol or confusing data interpretation.
* Subject has clinical conditions such as heart diseases, difficult-to-control blood pressure, difficult-to-control insulin-dependent diabetes or serious prior infections attributed to the diabetes, or others that, at the investigator's discretion, could seriously affect the subject's current clinical condition during study procedures.
* Subject has previous participation in the DETECT Study, current participation or previous participation in another drug or device study in the past 30 days that conflicts with this study as determined by the study sponsor.
* Subject has experienced gastro-intestinal hemorrhage in the past 6 months.
* Subject has any situation in which the use of aspirin is contraindicated for at least 6 months.
* Subject has epilepsy.
* Subject has known severe allergies, e.g., peanut, bee sting, etc.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1020 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2014-05-01 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
The primary efficacy objective is to determine that the Guardian System reduces the composite of Cardiac or unexplained death, new Q-wave MI and time to door for a confirmed occlusive event at a medical facility >2 hours. | Due to Bayesian statistical analysis, the study data will be analyzed after subject enrollment reaches 600, 900, 1200, etc. With amendment the study period spanned from December 2008 until database lock April 1, 2014.
  With Amendment the primary efficacy objective was amended to be a co-primary endpoint which included A) a hypothesis test of superiority for positive predictive value of ER visits in the ALARMS_ON group due to Guardian alerting (with or without concurrent symptoms) compared to ER visits in the ALARMS_OFF group due to symptoms only; AND B) a hypothesis test of non-inferiority for rate of false positive ER visits in the ALARMS_ON group due to Guardian alerting (with or without concurrent symptoms) compared to rate of false positive ER visits in the ALARMS_OFF group due to symptoms only.

SECONDARY OUTCOMES:
- Reduction of the incidence of cardiac death or unexplained death during follow-up - Reduction of the incidence of "New" Q-wave myocardial infarction in one or more distributions during follow-up- Reduction of the time to door for confirmed STEMI. | Due to Bayesian statistical analysis, the study data will be analyzed after subject enrollment reaches 600, 900, 1200, etc With amendment the study period spanned from December 2008 until database lock April 1, 2014.
  With Amendment the secondary efficacy endpoint measures were amended to include Endpoint #1) a hypothesis test of superiority for rate of false positive ER visits in the ALARMS_ON group due to Guardian alerting (with or without concurrent symptoms) compared to rate of false positive ER visits in the ALARMS_OFF group due to symptoms only.
Secondary Endpoint #2 | With amendment the study period spanned from December 2008 until database lock April 1, 2014.
  With Amendment the secondary efficacy endpoint measures were amended to include Endpoint #2) The number of Silent MIs, the percentage in relation to total MIs in the ALARMS ON group, and the percentage of subjects experiencing Silent MIs will be reported (no hypotheses existed for this endpoint)
Secondary Endpoint #3 | With amendment the study period spanned from December 2008 until database lock April 1, 2014.
  With Amendment the secondary efficacy endpoint measures were amended to include Endpoint #3) Descriptive statistics for the median, average and distribution of symptom-to-door and alarm-to-door times for STEMI events and the number and percentage of subjects with time-to-door times of < 2 hours will be reported for both the ALARMS ON and ALARMS OFF groups (no hypotheses existed for this endpoint).
Secondary Endpoint #4 | With amendment the study period spanned from December 2008 until database lock April 1, 2014.
  With Amendment the secondary efficacy endpoint measures were amended to include Endpoint #4) The time that elapses between the initial patient prompt (alarm or symptom) and arrival at a medical facility will be calculated for all subjects who suffered a STEMI or NSTEMI, and had an associated Guardian alarm (no hypotheses existed for this endpoint).
Secondary Endpoint #5 | With amendment the study period spanned from December 2008 until database lock April 1, 2014.
  With Amendment the secondary efficacy endpoint measures were amended to include Endpoint #5: The time that elapses between the initial patient prompt (Alarm or Symptom) and arrival at a medical facility will be calculated for all subjects who suffered an ACS event (STEMI, NSTEMI, or Unstable Angina), and had an associated Guardian System alarm (with or without symptoms) (no hypotheses existed for this endpoint).

CONTACTS AND LOCATIONS:
Locations (94):
- United States (94):
  - Cardiology, P.C., Birmingham, Alabama
  - Heart Center Research/Huntsville Hospital, Huntsville, Alabama
  - Banner Heart Hospital, Mesa, Arizona
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Southwest Heart Group, Tucson, Arizona
  - John Muir Clinical Research Center, Concord, California
  - California Clinical Research Foundation, Glendale, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Mission Internal Medical Group, Mission Viejo, California
  - Orange County Heart Institute and Research Center Hospital, Orange, California
  - Huntington Memorial Hospital, Pasadena, California
  - University of California Davis Medical Center, Sacramento, California
  - Sutter Memorial Hospital, Sacramento, California
  - Salinas Valley Memorial Hospital, Salinas, California
  - Radiant Research, Santa Rosa, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - Daytona Heart Group, Daytona Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - NorthFL/South GA VA Health System, Gainesville, Florida
  - Mercy Research Institute, Miami, Florida
  - University of Miami, Miami, Florida
  - New Phase Clinical Trials, Miami Beach, Florida
  - Complete Cardiology Care, New Smyrna Beach, Florida
  - East Coast Institute for Research, Saint Augustine, Florida
  - Univeristy of South Florida, Tampa, Florida
  - Florida Hospital - Pepin Heart Institute, Tampa, Florida
  - The Medical Center of Central Georgia, Macon, Georgia
  - Northwestern University, Chicago, Illinois
  - Advocate Medical Group, Park Ridge, Illinois
  - Premier Healthcare, Bloomington, Indiana
  - Northern Indiana Research Alliance, Fort Wayne, Indiana
  - Heart Center of Lake County, Merrillville, Indiana
  - Medical Consultants, PC, Muncie, Indiana
  - Central Baptist Hospital, Lexington, Kentucky
  - Innovative Medical Research, Covington, Louisiana
  - Heart Clinic of Hammond, Hammond, Louisiana
  - Louisiana Heart Center, Slidell, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - MedStar Health Research Institute, Baltimore, Maryland
  - Suburban Hospital - Johns Hopkins Medicine, Bethesda, Maryland
  - Woodholme Cardiovacular Associates, Pikesville, Maryland
  - Washington Adventist Hospital, Takoma Park, Maryland
  - McLaren Bay Region, Bay City, Michigan
  - DMC Cardiovascular Institute at Harper-Hutzel Hospital, Detroit, Michigan
  - Detroit Clinical Research Center, Farmington Hills, Michigan
  - Cardiology Consultants of East Michigan, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - McLaren Macomb, Mount Clemens, Michigan
  - Cardiac & Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - University of Medicine & Dentistry NJ, New Brunswick, New Jersey
  - St. Michael's Medical Center, Newark, New Jersey
  - Lourdes Cardiology Services, Voorhees Township, New Jersey
  - Albany Associates in Cardiology, Albany, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Buffalo Heart Group - Mercy Hospital of Buffalo, Buffalo, New York
  - Buffalo Heart Group - Millard Fillmore Gates Circle Hospital, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Cardiology Group of Western New York, Williamsville, New York
  - REX Healthcare, Raleigh, North Carolina
  - Good Samaritan Hospital, Dayton, Ohio
  - Cardiovascular Research Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - South Oklahoma Heart Research, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - St. Mary Medical Center Research Institute, Langhorne, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - Donald Guthrie Foundation for Education & Research, Sayre, Pennsylvania
  - Geisinger Wyoming Valley Heart Hospital, Wilkes-Barre, Pennsylvania
  - Cardiac Diagnostic Associates/York Hospital, York, Pennsylvania
  - AnMed Health, Anderson, South Carolina
  - Greenville Hospital System, Greenville, South Carolina
  - Stern Cardiovascular Center, Germantown, Tennessee
  - Turkey Creek Medical Center, Knoxville, Tennessee
  - St. Thomas Research Institute, Nashville, Tennessee
  - Cardiology Center of Amarillo, Amarillo, Texas
  - West Houston Area Clinical Trial Consultants, Houston, Texas
  - Scott and White Healthcare, Temple, Texas
  - Tyler Cardiovascular Consultants, Tyler, Texas
  - Cardiology Associates of Fredericksburg, Fredericksburg, Virginia
  - Virginia Cardiovascular Associates, Manassas, Virginia
  - Riverside Regional Medical Center, Newport News, Virginia
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Cardiovascular Associates, Ltd, Virginia Beach, Virginia
  - Swedish Medical Center/Cardiovascular Research, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
When we have completed review with the FDA, the IPD will will be made available.

REFERENCES:
- [Derived] Holmes DR Jr, Krucoff MW, Mullin C, Mikdadi G, Presser D, Wohns D, Kaplan A, Ciuffo A, Eberly AL 3rd, Iteld B, Fischell DR, Fischell T, Keenan D, John MS, Gibson CM. Implanted Monitor Alerting to Reduce Treatment Delay in Patients With Acute Coronary Syndrome Events. J Am Coll Cardiol. 2019 Oct 22;74(16):2047-2055. doi: 10.1016/j.jacc.2019.07.084. PMID 31623762
- [Derived] Gibson CM, Holmes D, Mikdadi G, Presser D, Wohns D, Yee MK, Kaplan A, Ciuffo A, Eberly AL 3rd, Iteld B, Krucoff MW. Implantable Cardiac Alert System for Early Recognition of ST-Segment Elevation Myocardial Infarction. J Am Coll Cardiol. 2019 Apr 23;73(15):1919-1927. doi: 10.1016/j.jacc.2019.01.014. Epub 2019 Mar 3. PMID 30842028
- [Derived] Rogers T, Steinvil A, Torguson R, Waksman R. Overview of the 2016 US Food and Drug Administration Circulatory System Devices Panel Meeting on the AngelMed Guardian System. Circulation. 2016 Jul 19;134(3):262-4. doi: 10.1161/CIRCULATIONAHA.116.023081. No abstract available. PMID 27436882
- [Derived] Gibson MC, Krucoff M, Fischell D, Fischell TA, Keenan D, Abueg C, Patel C, Holmes D. Rationale and design of the AngeLmed for Early Recognition and Treatment of STEMI trial: a randomized, prospective clinical investigation. Am Heart J. 2014 Aug;168(2):168-74. doi: 10.1016/j.ahj.2014.05.008. Epub 2014 May 24. PMID 25066555